CLINICAL TRIAL: NCT01697631
Title: Comparison of Biphasic Insulin Aspart 30 Twice Daily and Biphasic Insulin Aspart 30 Twice Daily Plus Lunchtime Injection of Insulin Aspart Treatment Efficiency in Overall Glycemic Control and Postprandial Glycemic Excursions. A Multi-center, Randomized, Open-label, Two-armed Parallel Group Trial in Subjects With Type 2 Diabetes Previously Treated With Conventional Biphasic Human Insulin 30/70
Brief Title: Glycemic Control of Biphasic Insulin Aspart 30 in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1409
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp (Experimental)
  Interventions: Drug: biphasic insulin aspart 30
- Insulin aspart (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: insulin aspart

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Administrated subcutaneously (s.c., under the skin) at breakfast and evening main meals
Drug: insulin aspart — Administrated subcutaneously (s.c., under the skin) before lunch
  Arms: Insulin aspart

SUMMARY:
This this trial is conducted in Europe. The aim of this trial is to compare glycaemic control of biphasic insulin aspart 30 (BIAsp 30) alone or combined with insulin aspart(IAsp) in patients previously treated with conventional Biphasic Human Insulin 30/70.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Current treatment with conventional biphasic human insulin 30/70 b.i.d. (twice daily) for at least 3 months
* HbA1c (glycosylated haemoglobin) equal to or below 12%
* Willing and able to perform self blood glucose monitoring (SMBG)

Exclusion Criteria:

* History of drug or alcohol dependence
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation
* Previous participation in this trial
* Receipt of any investigational drug within the last month prior to this trial
* Known or suspected allergy to trial products or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2002-07-22 (Actual); Primary Completion 2003-04-24 (Actual); Study Completion 2003-04-24 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
7-point blood glucose profile
Correlation of endpoint HbA1c with baseline BMI (body mass index) and HbA1c with treatment mode stratification
Incidence of adverse events
Hypoglycaemic episodes (minor, major or nocturnal)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (12):
- Poland (12):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Bytom
  - Novo Nordisk Investigational Site, Kamieniec Ząbkowicki
  - Novo Nordisk Investigational Site, Katowice
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Nysa
  - Novo Nordisk Investigational Site, Otwock
  - Novo Nordisk Investigational Site, Radom
  - Novo Nordisk Investigational Site, Ruda Śląska
  - Novo Nordisk Investigational Site, Sosnowiec
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com